CLINICAL TRIAL: NCT05219799
Title: Sex Disparities in Hypoxic Vasodilation and Impact of Obesity
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Assistant Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2080504
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Vasodilation; Healthy
MeSH Terms: conditions — Obesity; Aneurysm | interventions — Propranolol; Isoproterenol; Phentolamine; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypoxia Exposure (Other): Men and women will be exposed to isocapnic hypoxia. Participants will wear a mask and systemic oxygen levels will be titrated to attain hypoxemia as assessed by pulse oximetry.
  Interventions: Drug: Propranolol Hydrochloride; Drug: Isoproterenol; Drug: Phentolamine Mesylate; Drug: Norepinephrine

INTERVENTIONS:
Drug: Propranolol Hydrochloride — Regional forearm blockade of β-adrenergic receptors at 20 mcg/dL/min via brachial artery catheter during normoxia and hypoxia exposures
Drug: Isoproterenol — Dose response (1, 3, 6, and 12 ng/dL/min) regional infusion to assess β-adrenergic receptor responsiveness
Drug: Phentolamine Mesylate — This infusion will be for 10 min before baseline measurement (12 mcg/dL/min) and continue the infusion at a maintenance rate (5 mcg/dL/min).
Drug: Norepinephrine — Regional forearm infusion at 8 ng/dL/min via brachial artery catheter during normoxia and hypoxia exposures

SUMMARY:
The purpose of this project is to examine key mechanisms contributing to sex-differences in hypoxic vasodilation and the impact of obesity, with particular emphasis on the sympathetic nervous system.

DETAILED DESCRIPTION:
Patients with sleep apnea are at increased risk of developing cardiovascular disease - with women at potentially greater risk than men. Contributing mechanisms are not well understood, but may be related to how women respond to low oxygen and, given over 70% of patients with sleep apnea are obese, the impact of obesity. This project seeks to increase our understanding of mechanisms that may contribute to sex differences in the cardiovascular response to low oxygen with the hope that this knowledge will improve the efficacy of current therapies and support the discovery of novel therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* BMI >18 kg/m2

Exclusion Criteria:

* Pregnancy, breastfeeding
* Diagnosed sleep apnea or AHI >10 events/hr
* Current smoking/Nicotine use
* Increased risk of bleeding, pro-coagulant disorders, clotting disorders, anticoagulation therapy
* Nerve/neurologic disease
* Cardiovascular, hepatic, renal, respiratory disease
* Blood pressure ≥140/90 mmHg
* Diabetes, Polycystic ovarian syndrome
* Communication barriers
* Prescription medications, Sensitivity to lidocaine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in forearm vascular conductance with intra-arterial drug infusion | Change from baseline to last 1-minute of drug infusion
  Vascular conductance is an index of vascular tone and is measured using a technique called venous occlusion plethysmography.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Limberg, Ph.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided